CLINICAL TRIAL: NCT01837641
Title: A Single-Dose and Multiple-Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY3002813 in Patients With Mild Cognitive Impairment Due to Alzheimer's Disease or Mild to Moderate Alzheimer's Disease
Brief Title: A Study of LY3002813 in Participants With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15082; I5T-MC-AACC (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- LY3002813-Single 0.1 mg/kg then multiple 0.3 mg/kg (Experimental): 0.1 milligram per kilogram (mg/kg) single dose then 0.3 mg/kg LY3002813 given every 4 weeks for up to 16 weeks intravenously (IV)
  Interventions: Biological: LY3002813-IV
- LY3002813-Single then multiple 0.3 mg/kg (Experimental): 0.3 mg/kg single dose then 0.3 mg/kg LY3002813 given every 4 weeks for up to 16 weeks IV
  Interventions: Biological: LY3002813-IV
- LY3002813-Single 1 mg/kg in Healthy Participants (Experimental): 1 mg/kg single dose LY3002813 given once by IV infusion.
  Interventions: Biological: LY3002813-IV
- LY3002813-Single then multiple 1 mg/kg (Experimental): 1 mg/kg single dose then 1 mg/kg LY3002813 given every 4 weeks for up to 16 weeks IV
  Interventions: Biological: LY3002813-IV
- LY3002813-Single then multiple 3 mg/kg (Experimental): 3 mg/kg single dose then 3 mg/kg LY3002813 given every 4 weeks for up to 16 weeks IV
  Interventions: Biological: LY3002813-IV
- LY3002813-Single then multiple 10 mg/kg (Experimental): 10 mg/kg single dose then 10 mg/kg LY3002813 given every 4 weeks for up to 16 weeks IV
  Interventions: Biological: LY3002813-IV
- Placebo-Single then multiple (Placebo Comparator): Placebo given once, then every 4 weeks for up to 16 weeks IV
  Interventions: Drug: Placebo-IV
- LY3002813-SC (Experimental): Up to 3 mg/kg LY3002813 given once subcutaneously (SC)
  Interventions: Biological: LY3002813-SC
- LY3002813-IV (Experimental): Up to 3mg/kg LY3002813 given once intravenously (IV)
  Interventions: Biological: LY3002813-IV

INTERVENTIONS:
Biological: LY3002813-IV — Administered IV
  Arms: LY3002813-IV; LY3002813-Single 0.1 mg/kg then multiple 0.3 mg/kg; LY3002813-Single 1 mg/kg in Healthy Participants; LY3002813-Single then multiple 0.3 mg/kg; LY3002813-Single then multiple 1 mg/kg; LY3002813-Single then multiple 10 mg/kg; LY3002813-Single then multiple 3 mg/kg
Biological: LY3002813-SC — Administered SC
  Arms: LY3002813-SC
Drug: Placebo-IV — Administered IV
  Arms: Placebo-Single then multiple

SUMMARY:
The study will evaluate the safety of LY3002813 by looking at adverse events. The study will also look at the effect the body has on LY3002813. Study participants will be healthy or will have mild cognitive impairment (MCI) due to Alzheimer's disease (AD) or mild to moderate AD.

There will be seven groups of study participants. Five groups will receive a single dose of LY3002813 or placebo (no drug), followed by up to 4 multiple doses of LY3002813 or placebo given as an injection into a vein. Approximately 12 weeks will pass between the single dose and the first multiple dose. One group of participants will receive a single dose of LY3002813 given as an injection under the skin. One group of participants will receive a single dose of LY3002813 given as an injection into a vein.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Participants:

  * Overtly healthy males, as determined by medical history and physical examination, willing to use a reliable method of birth control and will not donate sperm during the study
  * Between 18 to 40 years old.
  * Body Mass Index (BMI) of between 18.0 and 30.0 kilogram per meter square (kg/m^2), inclusive
* Participants with Mild Cognitive Impairment Due to Alzheimer's Disease (AD) or AD:

  * Present with mild cognitive impairment (MCI) due to AD or mild-to-moderate AD
  * Men or nonfertile women, at least 50 years of age. Nonfertile is defined as hysterectomy and/or bilateral oophorectomy, or amenorrhea for at least 1 year
  * Have a caregiver/study informant who provides a separate written informed consent to participate
  * Have adequate vision and hearing for neuropsychological testing in the opinion of the investigator
  * Positive florbetapir scan

Exclusion Criteria:

-Healthy Participants: Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, immunological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data

* Participants with Mild Cognitive Impairment Due to AD or AD:

  * Do not have a reliable caregiver/study informant who is in frequent contact with the participant, who will accompany the participant to the office and/or be available by telephone at designated times, and will monitor administration of prescribed medications
  * Are being monitored for radiation due to occupational exposure to ionized radiation, or exposure to ionizing radiation within last 12 months from an investigational study
  * History within the past 5 years of a primary or recurrent malignant disease with the exception of resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or in situ prostate cancer with a normal prostate-specific antigen post resection
* All Participants:

  * History of intracranial hemorrhage, cerebrovascular aneurysm or arteriovenous malformation, or carotid artery occlusion, or stroke or epilepsy
  * Have any contraindications for magnetic resonance imaging (MRI) studies, including claustrophobia, the presence of contraindicated metal (ferromagnetic) implants, cardiac pacemaker
  * Have allergies to humanized monoclonal antibodies, including proteins and diphenhydramine, epinephrine, and methylprednisolone
  * Have gamma globulin therapy within the last year
  * Previously dosed in any other study investigating active immunization against amyloid beta (Aβ)
  * Previously dosed in any other study investigating passive immunization against Aβ within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-05-03 (Actual); Primary Completion 2016-08-24 (Actual); Study Completion 2016-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (4):
  - Collaborative Neuroscience Network - CNS, Long Beach, California
  - Compass Research, Orlando, Florida
  - Atlanta Center of Medical Research, Atlanta, Georgia
  - PRAHealthSciences, Salt Lake City, Utah
- Japan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sumida-Ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Dose-escalation study in participants(pts) with mild cognitive impairment (MCI) due to Alzheimer's disease (AD).Under an amendment,Pharmacokinetics of unblinded single IV dose of 1 milligram per kilogram (mg/kg) LY3002813 in young,healthy male pts was assessed if absence of amyloid target affected the PK as compared to amyloid-positive pts with AD.
Groups:
- Placebo IV: Single dose of placebo matching LY3002813 given once, then every 4 weeks for up to 16 weeks by intravenous (IV) infusion.
- 0.1 mg/kg / 0.3 mg/kg LY3002813 IV: Single dose of 0.1 milligram per kilogram (mg/kg) LY3002813 given once, then 0.3 mg/kg LY3002813 every 4 weeks for up to 16 weeks by IV infusion.
- 0.3 mg/kg LY3002813 IV: Single dose of 0.3 mg/kg LY3002813 given once, then every 4 weeks for up to 16 weeks by IV infusion.
- 1 mg/kg LY3002813 IV: Healthy Participants: Single dose of 1 mg/kg LY3002813 given once by IV infusion.
- 1 mg/kg LY3002813 IV: Single dose of 1 mg/kg LY3002813 given once, then every 4 weeks for up to 16 weeks by IV infusion.
- 3 mg/kg LY3002813 IV: Single dose of 3 mg/kg LY3002813 given once, then every 4 weeks for up to 16 weeks by IV infusion.
- 10 mg/kg LY3002813 IV: Single dose of 10 mg/kg LY3002813 given once, then every 4 weeks for up to 16 weeks by IV infusion.
- 3 mg/kg LY3002813 SC: Single dose of 3 mg/kg LY3002813 given once subcutaneously (SC).
Period: Overall Study
Arm/Group | Placebo IV | 0.1 mg/kg / 0.3 mg/kg LY3002813 IV | 0.3 mg/kg LY3002813 IV | 1 mg/kg LY3002813 IV: Healthy Participants | 1 mg/kg LY3002813 IV | 3 mg/kg LY3002813 IV | 10 mg/kg LY3002813 IV | 3 mg/kg LY3002813 SC
Started | 12 | 4 | 7 | 6 | 9 | 11 | 6 | 8
Received at Least 1 Dose of Study Drug | 12 | 4 | 7 | 6 | 9 | 11 | 6 | 8
Completed | 11 | 4 | 7 | 6 | 8 | 9 | 5 | 8
Not Completed | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Not completed — Sponsor decision | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug.
Groups:
- Placebo IV: Single dose of placebo matching LY3002813 given once, then every 4 weeks for up to 16 weeks by IV infusion.
- 0.1 mg/kg / 0.3 mg/kg LY3002813 IV: Single dose of 0.1 mg/kg LY3002813 given once, then 0.3 mg/kg LY3002813 every 4 weeks for up to 16 weeks by IV infusion.
- 3 mg/kg LY3002813 SC: Single dose of 3 mg/kg LY3002813 given once SC.
- Total: Total of all reporting groups
Arm/Group | Placebo IV | 0.1 mg/kg / 0.3 mg/kg LY3002813 IV | 0.3 mg/kg LY3002813 IV | 1 mg/kg LY3002813 IV: Healthy Participants | 1 mg/kg LY3002813 IV | 3 mg/kg LY3002813 IV | 10 mg/kg LY3002813 IV | 3 mg/kg LY3002813 SC | Total
Number analyzed (Participants) | 12 | 4 | 7 | 6 | 9 | 11 | 6 | 8 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.8 (4.9) | 71.3 (11.6) | 75.0 (8.4) | 25.8 (3.3) | 74.7 (9.3) | 73.0 (8.8) | 72.3 (10.7) | 74.5 (9.5) | 69.7 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 4 | 0 | 4 | 8 | 2 | 5 | 33
  Male | 5 | 1 | 3 | 6 | 5 | 3 | 4 | 3 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 4
  Not Hispanic or Latino | 12 | 4 | 7 | 4 | 8 | 11 | 5 | 8 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 2 | 3 | 0 | 3 | 4 | 2 | 2 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3
  White | 6 | 2 | 3 | 5 | 6 | 6 | 4 | 6 | 38
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 2 | 4 | 6 | 6 | 7 | 4 | 6 | 43
  Japan | 4 | 2 | 3 | 0 | 3 | 4 | 2 | 2 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Events (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: Data presented are the number of participants who experienced SAEs which were considered to be related to study treatment by the investigator while on treatment and during the follow-up. Summaries of SAEs and other non-serious adverse events (AEs), regardless of causality, are located in the Reported Adverse Events module.
Time Frame: Day 1 up to Day 253
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV | 0.1 mg/kg / 0.3 mg/kg LY3002813 IV | 0.3 mg/kg LY3002813 IV | 1 mg/kg LY3002813 IV: Healthy Participants | 1 mg/kg LY3002813 IV | 3 mg/kg LY3002813 IV | 10 mg/kg LY3002813 IV | 3 mg/kg LY3002813 SC
Number analyzed (Participants) | 12 | 4 | 7 | 6 | 9 | 11 | 6 | 8
Participants | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY3002813
Description: Maximum Concentration (Cmax) of LY3002813 after the first dose was evaluated.
Time Frame: Pre-dose, end of infusion for IV or 1h post injection for SC, 3, 24, 72, 96(SC), 120(SC), 144(SC), 168, 336, 504, 672, 1008, 1344, 1680 and 2016 hours (h) post-dose
Population: All enrolled participants who received at least 1 dose of study drug and have evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | 0.1 mg/kg / 0.3 mg/kg LY3002813 IV | 0.3 mg/kg LY3002813 IV | 1 mg/kg LY3002813 IV: Healthy Participants | 1 mg/kg LY3002813 IV | 3 mg/kg LY3002813 IV | 10 mg/kg LY3002813 IV | 3 mg/kg LY3002813 SC
Number analyzed (Participants) | 4 | 7 | 6 | 9 | 11 | 6 | 8
microgram per milliliter (μg/mL) | 2.90 (35) | 5.99 (77) | 31.5 (29) | 21.7 (21) | 71.6 (24) | 218 (16) | 12.0 (34)

3. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Time Zero to Infinity [AUC(0-∞)] of LY3002813
Description: Area Under the Concentration Versus Time Curve From Time Zero to Infinity [AUC(0-∞)] of LY3002813 after the first dose was evaluated.
Time Frame: Pre-dose, end of infusion for IV or 1h post injection for SC, 3, 24, 72, 96(SC), 120(SC), 144(SC), 168, 336, 504, 672, 1008, 1344, 1680 and 2016h post-dose
Population: All enrolled participants who received at least 1 dose of study drug and have evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day per milliliter (μg*day/mL)
Arm/Group | 0.1 mg/kg / 0.3 mg/kg LY3002813 IV | 0.3 mg/kg LY3002813 IV | 1 mg/kg LY3002813 IV: Healthy Participants | 1 mg/kg LY3002813 IV | 3 mg/kg LY3002813 IV | 10 mg/kg LY3002813 IV | 3 mg/kg LY3002813 SC
Number analyzed (Participants) | 4 | 7 | 6 | 9 | 11 | 6 | 8
microgram*day per milliliter (μg*day/mL) | 7.94 (32) | 26.3 (33) | 91.6 (17) | 79.9 (26) | 263 (19) | 1140 (39) | 157 (41)

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 253
Description: All enrolled participants who received at least 1 dose of study drug.
Arm/Group | Placebo IV | 0.1 mg/kg / 0.3 mg/kg LY3002813 IV | 0.3 mg/kg LY3002813 IV | 1 mg/kg LY3002813 IV: Healthy Participants | 1 mg/kg LY3002813 IV | 3 mg/kg LY3002813 IV | 10 mg/kg LY3002813 IV | 3 mg/kg LY3002813 SC
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/4 | 2/7 | 0/6 | 1/9 | 0/11 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 8/12 | 3/4 | 4/7 | 3/6 | 6/9 | 7/11 | 2/6 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo IV (N=12) | 0.1 mg/kg / 0.3 mg/kg LY3002813 IV (N=4) | 0.3 mg/kg LY3002813 IV (N=7) | 1 mg/kg LY3002813 IV: Healthy Participants (N=6) | 1 mg/kg LY3002813 IV (N=9) | 3 mg/kg LY3002813 IV (N=11) | 10 mg/kg LY3002813 IV (N=6) | 3 mg/kg LY3002813 SC (N=8)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo IV (N=12) | 0.1 mg/kg / 0.3 mg/kg LY3002813 IV (N=4) | 0.3 mg/kg LY3002813 IV (N=7) | 1 mg/kg LY3002813 IV: Healthy Participants (N=6) | 1 mg/kg LY3002813 IV (N=9) | 3 mg/kg LY3002813 IV (N=11) | 10 mg/kg LY3002813 IV (N=6) | 3 mg/kg LY3002813 SC (N=8)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral lichen planus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (5) | 3 (8) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral microhaemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Apathy (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Persecutory delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micrographic skin surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less